CLINICAL TRIAL: NCT01605305
Title: Phase II Study on FOLFOX6 as First-line Therapy to Treat Recurrent or Metastatic Esophageal Cancer
Brief Title: Study on FOLFOX6 as First-line Therapy to Treat Recurrent or Metastatic Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chang Jian Hua, associate chief physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: FOLFOX6-2008
Record Dates: First submitted 2012-05-22; First posted 2012-05-24 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Folfox protocol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFOX6 (Experimental)
  Interventions: Drug: FOLFOX6

INTERVENTIONS:
Drug: FOLFOX6 — OXA 100mg/m2 ivgtt 2h d1 LV 400mg/m2 ivgtt 2h d1 5FU 400mg/m2 iv. d1 5FU 2.4g/m2 civ 46h

SUMMARY:
The aim of this study is to explore whether FOLFOX6 as treatment could improve the time to progression (TTP) and overall survival (OS) of the patient with recurrent or metastatic esophagus.

DETAILED DESCRIPTION:
Explore whether FOLFOX6 as treatment could improve the TTP and OS of the patient with recurrent or metastatic esophagus

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven primary thoracic esophageal squamous cell carcinoma
2. Without chemotherapy or neo-adjuvant chemotherapy in 6 weeks ,radiotherapy has end at least 1 month,target lesion was not in an irradiated area.
3. Presence of at least one index lesion measurable by CT scan or MRI
4. 18~75 years
5. kps ≥ 70
6. Life expectancy of ≥ 3 months
7. ANC ≥ 2×109/L，PLT ≥ 100×109/L，Hb ≥ 90g/L
8. Cr ≤ 1.0×UNL
9. TB ≤ 1.25×UNL； ALT/AST ≤ 2.5×UNL，THE patient with liver metastasis ALT/AST ≤ 5.0×UNL；AKP ≤ 2.5×UNL
10. Signed written informed consent

Exclusion Criteria:

1. Previous exposure to oxa therapy in one year
2. diameter of tumor abdominal ≥ 10cm, Total volumes of liver lesions ≥ 50%,lung metastasis ≥ 25% total lung
3. chronic diarrhea,enteritis,intestine obstruction which are not under control
4. Psychiatric or addictive disorders that preclude obtaining informed consent or adherence to protocol.
5. peripheral neuropathy ≥ CTCAE 1
6. Other serious disease
7. Previous or concomitant malignancies except non-melanoma skin cancer, carcinoma in situ of the cervix, and invasive carcinoma of the colon, thyroid, cervix, or endometrium treated five years prior to study entry.
8. USE OTHER ANTITUMOR THERAPY
9. Breast-feeding or pregnant women, no effective contraception if risk of conception exists

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
TPP | from the first cycle of treatment (day one) to two month after the last cycle

SECONDARY OUTCOMES:
OS | from the first cycle of treatment (day one) to two month after the last cycle

CONTACTS AND LOCATIONS:
Overall Officials: chang j h, post-doctor, Principal Investigator — Fudan University